CLINICAL TRIAL: NCT01264835
Title: Assessment of a Slotted Anoscope That Facilitates Hemorrhoidectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-10-0003
Record Dates: First submitted 2010-12-17; First posted 2010-12-22 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Excisional Hemorrhoidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Slotted Anoscope — SA411

SUMMARY:
This trial is designed to assess intra-operative procedure outcomes (e.g.,procedure duration) and post-operative patient outcomes (e.g., pain)following a modified Ferguson hemorrhoidectomy procedure using the Slotted Anoscope with Harmonic or monopolar energy.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age
* Are willing to give consent and comply with evaluation and treatment schedule
* Meet institutional criteria for excisional hemorrhoidectomy
* Are able to understand and complete study questionnaires.

Exclusion Criteria:

* Previous Hemorrhoid surgery
* Chronic daily narcotic use
* Chronic Nonsteroidal Anti-inflammatory Drug use two weeks prior to procedure
* Internal hemorrhoids that may be suitable for office management (surgeon discretion)
* Fecal or urinary incontinence
* Inflammatory Bowel Disease (Crohns, ulcerative colitis)
* Acutely thrombosed hemorrhoids (surgeon discretion)
* Evidence of acute sepsis or the presence of a fistula
* Anal stricture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of South Alabama, Mobile, Alabama
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Slotted Anoscope: Subjects consenting to have hemorrhoidectomy with the slotted anoscope
Period: Overall Study
Arm/Group | Slotted Anoscope
Started | 2
Completed | 1
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Slotted Anoscope
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Procedure Duration (Surgery Time)
Description: Procedure duration was defined as the length of time in minutes from first insertion of the slotted anoscope to final removal of the slotted anoscope.
Time Frame: Time of surgery
Population: No analyses are being reported for this outcome measure as this trial was terminated early. The procedure was only performed with the slotted anoscope in 1 subject. No assessment or analysis of primary or secondary objectives was performed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Slotted Anoscope
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Slotted Anoscope
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Slotted Anoscope (N=2)
Rectal Ulceration (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No analyses are being reported for the primary outcome measure as this trial was terminated early. The procedure was only performed with the slotted anoscope in 1 subject. No assessment or analysis of primary or secondary objectives was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less